CLINICAL TRIAL: NCT02167581
Title: Confrontation Phenotypic (Clinical, Radiological, Histological) and Genotypic Epithelial Odontogenic Tumors Isolated or Syndromic Jaws
Brief Title: Confrontation Phenotypes and Genotypes of Epithelial Odontogenic Tumors of the Jaws
Acronym: TEIOS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081259
Record Dates: First submitted 2014-06-13; First posted 2014-06-19 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Epithelial Odontogenic Tumours
Keywords: Maxillofacial surgery; Epithelial odontogenic tumours

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — serum bank and tissue bank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- epithelial odontogenic tumours

SUMMARY:
Systematically compare the phenotype and genotype of epithelial odontogenic tumors in children and adults with a clinical, radiographic, pathologic and molecular level.

Either:

establish an observatory of this multidisciplinary tumor establish a tumor bank annotated scale unparalleled testing pathophysiological hypotheses search for prognostic factors.

DETAILED DESCRIPTION:
This is an observational study with retrospective and prospective parts. In retrospective part be included the Patients followed between 1992 and January 2011.

In prospective part will follow the Patients will be included after the starting of study.

There are 2 centers :

1. st center is in the service of Stomatology and Maxillofacial Surgery in the Pitie Salpetriere Hospital.
2. nd center is in the service of Maxillofacial Surgery in hospital Armand Trousseau.

Number of patients include in the part retrospective :

Center N°1-300adults Center N°2-90childrens

Number of patients include in the part prospective :

Center N°1- 90 Center N°2- 30

Duration of study is 3 years Duration of inclusion is 32 months Each patient will be followed for 4 months and for further up to 3 years from the first patient included.

We envision a next circuit : obtaining consent, preoperative consultation,surgery, postoperative consultation N°1, postoperative consultation N°2, genetics consultation and monitoring of patients in 6;12;18;24 months from surgery of tumor and limited in 3 years from th 1st patient included.

ELIGIBILITY:
Inclusion criteria

1. Patient with an osteolytic lesion of the jaws
2. Patient with epithelial odontogenic tumor:

   keratocysts ameloblastoma Pindborg tumor or calcifying (ESWT) Epidermoid (Squamous Odontogenic Tumor SOT) Clear cell (Clear Odontogenic Tumor Cells CCOT)
3. Patient monitoring in the period 1992 to January 2011 at the Trousseau Hospital (children) or at the Pitie Salpetriere (adult)
4. Patient aged 5 years or more
5. Adult patient who had signed informed consent
6. Holders of parental authority of minor patient were informed and signed consent

Non inclusion criteria

1. Patient with an osteolytic lesion of dental origin inflammatory (adjacent teeth decayed, non-living mortified)
2. Patient with a cyst fissure (nasopalatine, symphyseal or globulomaxillary)
3. Patient with arteriovenous malformation, vascular
4. Patient with cons-indication to MRI
5. Patient not affiliated with a social security scheme (beneficiary or assignee)
6. Pregnant woman
7. Patient in his history of hypersensitivity to salts of gadolinium
8. Patient receiving a measure of legal protection

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with an osteolytic lesion of the jaws resulting of an epithelial odontogenic tumor
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Phenotypic and genotypic lines connected to the epithelial odontogenic tumours | Month 24 from the surgery date
  In particular, to define the link between the genotype PTCH1, the size of the tumor, its osteolytic character and the predictive factors of recurrence.
  Data collection at M6, M12, M18, M24 from the surgery date

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Ruhin, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Stomatologie et Chirurgie Maxillofaciale - Pitie Salpetriere, Paris, France